CLINICAL TRIAL: NCT02983370
Title: Pilot Study for the Development of a Cortical Visual Neuroprosthesis for the Blind Based on Intracortical Microelectrodes
Brief Title: Development of a Cortical Visual Neuroprosthesis for the Blind
Acronym: CORTIVIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Hospital IMED Elche (Unknown)
Responsible Party: Principal Investigator, Eduardo Fernandez, MD and PhD, Universidad Miguel Hernandez de Elche
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CORTIVIS16-HUM1
Record Dates: First submitted 2016-09-12; First posted 2016-12-06 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Blindness
MeSH Terms: conditions — Blindness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blind volunteer (Experimental): Blind volunteers will be implanted with our existing vision neuroprosthetic system, which utilizes a FDA cleared microelectrode array, using a minicraniotomy. The array will be implanted near the occipital pole or in extra striate areas. The investigators will collect descriptive feedback regarding thresholds, evoked perceptions and stimulation parameters leading to recognizable patterns.
  Interventions: Procedure: Minicraniotomy

INTERVENTIONS:
Procedure: Minicraniotomy — The surgical method for the implantation of the intracortical microelectrodes is straightforward and follows the standard neurosurgical procedures. Briefly, after the scalp is prepped with an antiseptic, a small skin incision is made. Then the skin and muscles are lifted off from the bone and folded back. Next, one small burr hole or a minicraniotomy of approximately 1.5 cm is made in the skull. This is a minimally invasive procedure that allows an easy access to the brain and is a standard procedure widely used in neurosurgery.

SUMMARY:
The objective of this study is to evaluate the usefulness of a cortical visual prosthesis based on intracortical microelectrodes to provide a limited but useful sense of vision to profoundly blind. This pilot study will provide important information on safety and efficacy for the development of an useful cortical visual neuroprosthesis for the blind.

DETAILED DESCRIPTION:
Visual impairment is one of the ten most prevalent disabilities and poses extraordinary challenges to individuals in our society, which is heavily dependent on sight. Drug development and genetic engineering have had only marginal success as possible treatments but new hope has been generated by recent advances in neuroscience, micro-fabrication technologies, biomaterials, neuromorphic engineering and information and communication technologies leading to the development of highly sophisticated neural prosthetic devices which interact with the nervous system. Such assistive devices have already allowed thousands of deaf patients to hear sounds and acquire language abilities and the same hope exists in the field of visual rehabilitation.

Several research groups worldwide are engaged in attempts to restore vision through retinal prosthesis. However these devices are not viable for all causes of blindness. Thus, if the communication link between eye and brain is destroyed (e.g. for Glaucoma or optic nerve atrophy), as is the case for 148 million people worldwide, then visual cortical prosthesis holds the dominant hope for visual restoration. Consequently, there are many compelling reasons to pursue the development of a cortical prosthesis capable of restoring some useful vision in profoundly blind patients and this approach may be the only treatment available for end-stage retinitis pigmentosa patients and for pathologies such as glaucoma optic atrophy, trauma to the retina and/or optic nerves, and for diseases of the central visual pathways due to brain injuries or stroke.

The investigators will implant the CORTIVIS vision neuroprosthetic system, which utilizes a FDA cleared microelectrode array, into blind human volunteers and obtain descriptive feedback about visualized percepts. The experiments are designed to learn if volunteers can learn to integrate the electrical stimulation of brain visual areas into meaningful percepts. It is expected that a cortical device can create truly meaningful visual percepts that can be translated into functional gains such as the recognition, localization and grasping of objects or skillful navigation in familiar an unfamiliar environments resulting in a substantial improvement in the standard of living of blind and visually impaired persons.

All the experiments will be carried out at the patient's hospital room (Hospital IMED Elche) during the post-surgical period or in a human psychophysical laboratory (University Miguel Hernández).

ELIGIBILITY:
Inclusion Criteria:

* Participant is capable and willing to provide informed consent for participation in the trial.
* Severe visual impairment with bilateral visual loss.
* Greater than 18 years of age.
* General health: excellent.
* Following a general physical and neurological examination, patient must have normal serum electrolytes, C-reactive protein, complete blood count and PT and PTT.
* No history of stroke, seizure, coagulopathy, cardiac arrhythmias or ischemia, pulmonary, hepatic or renal disease, nor transmissible viruses such as hepatitis or HIV.
* Stable dose of current regular medication for at least four weeks prior to trial entry.
* Able to perform the study during the full time period of up to 6 months.

Special consideration will be given to patients with (1) detailed medical histories, including documentation of the onset, mechanism and evolution of the blindness; (2) lower risks associated with surgery; and (3) no psychiatric disorders or other mental disabilities.

Exclusion Criteria:

* Age <18 or >70.
* Period of appropriate visual functions < 12 years /lifetime.
* For medical reasons: Individuals with a history of seizure disorders, coagulopathy, cardiac arrythmias or ischemia, pulmonary, hepatic or renal disease, and any other neurological disorder. Patients who carry a transmissible virus such as hepatitis and individuals with HIV-related neuropathies.
* Vulnerable subject groups (e.g., pregnant women, prisoners, etc.).
* Persons unable to give written informed consent prior to participation in the study.
* Not able to perform the study during the full time period (at least 3 months).
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Thresholds of visual perceptions elicited by intracortical microstimulation | Within implantation period (up to 6 months)
  Charges needed for eliciting visual perceptions through electrical stimulation of the human cortex

SECONDARY OUTCOMES:
Phosphene mapping | Within implantation period (up to 6 months)
  Location of induced perceptions within the visual field by pointing with the finger where the phosphene is perceived
Visual Acuity | Within implantation period (up to 6 months)
  Spatial resolution measured by computerized visual tests
Motion perception | Within implantation period (up to 6 months)
  Correct perception of movement with a coarse pattern moving in one of four directions
Visual function | Within implantation period (up to 6 months)
  Effectiveness of intracortical microstimulation to recognize letters, habitual objects and complex stimulation patterrns as measured by a suite of visual function tests. Questionnaire.
Number of participants with significant adverse events. | Within implantation period (up to 6 months)
  Complications and adverse events will be assessed through participant description of any possible adverse event, neurological examination, clinical tests and a specific questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Fernandez, MD and PhD, Principal Investigator — Universidad Miguel Hernandez de Elche
Locations (2):
- Spain (2):
  - Hospital IMED Elche, Elche, Alicante
  - Universidad Miguel Hernandez de Elche, Elche, Alicante

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinez-Alvarez A, Crespo-Cano R, Diaz-Tahoces A, Cuenca-Asensi S, Ferrandez Vicente JM, Fernandez E. Automatic Tuning of a Retina Model for a Cortical Visual Neuroprosthesis Using a Multi-Objective Optimization Genetic Algorithm. Int J Neural Syst. 2016 Nov;26(7):1650021. doi: 10.1142/S0129065716500210. Epub 2016 Mar 29. PMID 27354187
- [Background] Alfaro A, Bernabeu A, Agullo C, Parra J, Fernandez E. Hearing colors: an example of brain plasticity. Front Syst Neurosci. 2015 Apr 14;9:56. doi: 10.3389/fnsys.2015.00056. eCollection 2015. PMID 25926778
- [Background] Fernandez E, Greger B, House PA, Aranda I, Botella C, Albisua J, Soto-Sanchez C, Alfaro A, Normann RA. Acute human brain responses to intracortical microelectrode arrays: challenges and future prospects. Front Neuroeng. 2014 Jul 21;7:24. doi: 10.3389/fneng.2014.00024. eCollection 2014. PMID 25100989
- [Background] Normann RA, Greger B, House P, Romero SF, Pelayo F, Fernandez E. Toward the development of a cortically based visual neuroprosthesis. J Neural Eng. 2009 Jun;6(3):035001. doi: 10.1088/1741-2560/6/3/035001. Epub 2009 May 20. PMID 19458403
- [Background] Warren DJ, Fernandez E, Normann RA. High-resolution two-dimensional spatial mapping of cat striate cortex using a 100-microelectrode array. Neuroscience. 2001;105(1):19-31. doi: 10.1016/s0306-4522(01)00174-9. PMID 11483297
- [Background] Maynard EM, Fernandez E, Normann RA. A technique to prevent dural adhesions to chronically implanted microelectrode arrays. J Neurosci Methods. 2000 Apr 15;97(2):93-101. doi: 10.1016/s0165-0270(00)00159-x. PMID 10788663
- [Background] Morillas CA, Romero SF, Martinez A, Pelayo FJ, Ros E, Fernandez E. A design framework to model retinas. Biosystems. 2007 Feb;87(2-3):156-63. doi: 10.1016/j.biosystems.2006.09.009. Epub 2006 Sep 7. PMID 17011701
- [Background] Fernandez E, Pelayo F, Romero S, Bongard M, Marin C, Alfaro A, Merabet L. Development of a cortical visual neuroprosthesis for the blind: the relevance of neuroplasticity. J Neural Eng. 2005 Dec;2(4):R1-12. doi: 10.1088/1741-2560/2/4/R01. Epub 2005 Nov 29. PMID 16317227
- [Background] Marin C, Fernandez E. Biocompatibility of intracortical microelectrodes: current status and future prospects. Front Neuroeng. 2010 May 28;3:8. doi: 10.3389/fneng.2010.00008. eCollection 2010. PMID 20577634
- [Background] Bernabeu A, Alfaro A, Garcia M, Fernandez E. Proton magnetic resonance spectroscopy (1H-MRS) reveals the presence of elevated myo-inositol in the occipital cortex of blind subjects. Neuroimage. 2009 Oct 1;47(4):1172-6. doi: 10.1016/j.neuroimage.2009.04.080. Epub 2009 May 5. PMID 19426816
- [Background] Normann RA, Fernandez E. Clinical applications of penetrating neural interfaces and Utah Electrode Array technologies. J Neural Eng. 2016 Dec;13(6):061003. doi: 10.1088/1741-2560/13/6/061003. Epub 2016 Oct 20. PMID 27762237
- [Background] Fernandez E, Alfaro A, Soto-Sanchez C, Gonzalez-Lopez P, Lozano AM, Pena S, Grima MD, Rodil A, Gomez B, Chen X, Roelfsema PR, Rolston JD, Davis TS, Normann RA. Visual percepts evoked with an intracortical 96-channel microelectrode array inserted in human occipital cortex. J Clin Invest. 2021 Dec 1;131(23):e151331. doi: 10.1172/JCI151331. PMID 34665780
- [Derived] Rocca A, Lehner C, Wafula-Wekesa E, Luna E, Fernandez-Cornejo V, Abarca-Olivas J, Soto-Sanchez C, Fernandez-Jover E, Gonzalez-Lopez P. Robot-assisted implantation of a microelectrode array in the occipital lobe as a visual prosthesis: technical note. J Neurosurg. 2023 Oct 27;140(4):1169-1176. doi: 10.3171/2023.8.JNS23772. Print 2024 Apr 1. PMID 37890180